CLINICAL TRIAL: NCT03315546
Title: Radiotherapy Delivery in Deep Inspiration for Pediatric Patients: TEDDI - a NOPHO Feasibility Study
Brief Title: Radiotherapy Delivery in Deep Inspiration for Pediatric Patients
Acronym: TEDDI
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Collaborators: Aarhus University Hospital (Other); Tampere University Hospital (Other); Helsinki University Central Hospital (Other)
Responsible Party: Principal Investigator, Maja Maraldo, Principal investigator, Rigshospitalet, Denmark
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-16035870
Record Dates: First submitted 2017-09-14; First posted 2017-10-20 (Actual); Last update posted 2020-10-09 (Actual); Status verified 2020-10

CONDITIONS: Pediatric Cancer
Keywords: deep inspiration breath-hold; radiotherapy; late effects; pediatric cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Intervention Model Description: non-randomised feasiblity study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Radiation: radiotherapy delivery in deep-inspiration — Radiotherapy delivery i deep-inspiration versus free-breathing

SUMMARY:
TEDDI is a non-randomised phase II trial in Scandinavia. All pediatric patients, referred for radiotherapy in the thorax or abdomen and irrespective of diagnosis, are eligible.

Deep inspiration breath-hold (DIBH) is a simple radiotherapy technique, which could have a dramatic impact on the risk of late effects in children. In DIBH, the radiotherapy is delivered while the patient holds his/her breath (4-6 sequential breath-holds). The anatomy is changed and imaging artifacts from respiratory movement are diminished. DIBH is widely used in adult patients with breast cancer and mediastinal lymphoma to minimize the risk of radiation-induced late effects due to a reduced dose to the healthy organs. Also, the technique is simple and cost-efficient.

For pediatric patients, the investigators aim to:

* Estimate the dosimetric benefit of radiotherapy using DIBH compared to free-breathing
* Establish the compliance of DIBH
* Determine if DIBH is an accurate and reproducible strategy
* Optimize treatment planning considering the risk from loss of tumour control as well as the risk of late effects.

DETAILED DESCRIPTION:
Background:

The majority (approximately 80%) of pediatric patients with cancer become long-term survivors. Long-term follow-up of childhood cancer survivors has documented a substantial treatment-induced increased mortality and morbidity, primarily from cardiovascular disease and second cancers. Specifically, cardiac mortality has been shown to be 5-fold higher, cardiac morbidity 2-fold to 6-fold higher, and the incidence of second cancers 8-fold higher in childhood cancer survivors compared to the general population or siblings. Due to the young age at diagnosis and corresponding long life expectancy of pediatric patients the impact of late effect(s) on patient quality of life, morbidity, and ultimately mortality is non-trivial.

Radiotherapy-induced late effects are severe, yet difficult to assess and quantify as they occur late and, therefore, often are the results of treatment regimens now considered outdated. Nonetheless, the risk of radiation-induced late effects is known to be influenced by both the radiation dose and the volume of irradiated tissue. In adults, the use of more conformal radiotherapy delivery techniques and breathing adaptation has been introduced in order to limit the irradiation of the surrounding healthy organs. However, there has been a reluctance to implement new radiotherapy delivery techniques in the treatment of pediatric patients as late effects data are not available for these new techniques and for the fear of a low compliance with breathing instructions.

Deep inspiration breath-hold (DIBH) is a simple radiotherapy technique, which could have a dramatic impact on late effects in children. In DIBH, the radiotherapy is delivered while the patient holds his/her breath (defined as 4 to 6 sequential breath-holds of ≥20 sec). In deep inspiration, the patient anatomy is changed and imaging artifacts from respiratory movement are diminished as the organs are not moving. Radiotherapy in DIBH can reduce the irradiation of the heart, breasts, and lungs without impacting the delivered radiation dose to the tumor and with no detriment to other healthy organs. Also, the technique is simple and cost-efficient. DIBH is widely used throughout the world in adult patients with left-sided breast cancer and with mediastinal lymphoma to minimize the risk of radiation-induced late effects.

The Department of Radiation Oncology at Rigshospitalet has pioneered the use of DIBH in the treatment of patients with breast cancer and mediastinal lymphoma [Korreman et al., Pedersen et al.] and is currently prospectively testing the DIBH technique in a more frail population of lung cancer patients. The department has extensive experience in the daily delivery and patient coaching of adult patients. While the experience from several centers confirms that the compliance of adult patients to DIBH is excellent, no reports exist of the applicability of DIBH to pediatric patients, especially the very young.

The investigators hypothesize that TEDDI is a feasible and reproducible strategy which will result in a 25% reduction in the mean radiation dose to the heart in pediatric patients referred for radiotherapy to tumors in the thorax or abdomen. This is expected to be true for all pediatric patients, regardless of age.

Through TEDDI, the investigators specifically aim to:

* Estimate the dosimetric benefit of radiotherapy using DIBH compared to free-breathing in pediatric patients.
* Establish the compliance of DIBH in pediatric patients in all age groups.
* Determine if DIBH is an accurate and reproducible strategy for pediatric patients.

Key research questions:

1. What is the extent of the dosimetric benefit of DIBH compared to free-breathing radiotherapy? For adult patients with breast cancer, malignant lymphoma, and lung cancer, radiotherapy delivered in DIBH compared to free-breathing significantly lowers the dose to the heart, lungs, and stomach. However, for very young patients the anatomical changes (i.e. inflation of the lungs, increased separation of the heart and the tumor) might be less pronounced than for adults hampering the dosimetric advantage of DIBH.

   Hypothesis 1 (H1): For more than 75% of patients, treatment in DIBH will be dosimetrically superior to treatment in free-breathing.
2. Is DIBH well tolerated by pediatric patients throughout their treatment? At present, the information material regarding DIBH and the visual feedback equipment (consisting of video goggles) is designed for and aimed at adult patients. In TEDDI, all aspects of the current DIBH workflow will be adapted in order to provide a comfortable setting for pediatric patients. Based on preliminary tests on healthy volunteers, children as young as 5 years are able to comply with the DIBH instructions given by the present visual feedback equipment.

   Hypothesis 2 (H2): over 90% of pediatric patients older than 5 years can perform a stable and comfortable DIBH (in the form of 4 to 6 sequential breath-holds of ≥20 sec) through their course of radiotherapy.
3. Can the prescribed radiation dose be delivered accurately and reproducibly to the tumor in DIBH? Interfraction monitoring will ensure reliable treatment between treatment days using the RPM system, and intrafraction monitoring will assess the stability of the patient positioning/breath-hold during the treatment. Image acquisition parameters will be optimized to provide sufficient image quality at the lowest possible radiation exposure.

Hypothesis 3 (H3): The tumor position will be reproducible from day to day, as well as from breath-hold to breath-hold. Variations in position will be less than 5 mm over the whole treatment course.

Treatment planning:

All diagnostic imaging during treatment and treatment planning will be performed according to national guidelines (as per cancer diagnosis). For the radiotherapy planning, a planning CT scan will be performed in DIBH as well as in free-breathing for each patient. On both scans the gross tumor volume (GTV), the clinical target volume (CTV) which comprises the GTV adjusted for normal tissue, and the planning target volume (PTV) which is the CTV including a planning margin, will be defined. All relevant, healthy organs at risk from radiation exposure will be contoured (e.g. heart, female breasts, lungs, esophagus, thyroid, salivary glands, spinal cord, bone marrow, stomach, spleen, kidneys, liver). A DIBH and a free-breathing radiotherapy plan will be calculated, both with similar planning objectives for the tumor and organs at risk. All DIBH treatment plans will be designed to keep the number of breath-holds per fraction as low as reasonably achievable (including image guidance) for patient comfort.

Whenever a PET scanning is considered an integral part of the radiotherapy planning, a PET scanning should also be performed in the treatment position in both DIBH and in free-breathing for optimal image fusion. However, for institutions where this is not feasible, participation in TEDDI is still possible.

Treatment delivery:

Patients will be treated in DIBH, if the calculated treatment plan in DIBH is superior to the treatment plan in free-breathing with respect to the lowest overall dose to the organs at risk while maintaining acceptable tumor coverage. Coverage of the CTV and PTV will have the highest priority, as per ICRU83 guidelines.

Follow-up:

Enrollment in TEDDI will not affect the standard follow-up program of pediatric patients which is diagnosis specific.

ELIGIBILITY:
Inclusion Criteria:

* Age 5-17 years.
* Patients with a tumor in the mediastinum or abdomen with possible need of radiotherapy according to current treatment guidelines, irrespective of cancer diagnosis.
* The ability to perform three sequential breath-holds of 20 seconds each during the coaching session.
* Written informed consent from parents or legal guardians.

Exclusion Criteria:

* Age younger than 5 years or older than 17 years.
* The need for radiotherapy under general anesthesia.
* CNS tumor or pelvic localization.
* Unable to understand coaching information directly or through interpretation.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
The dosimetric benefit of DIBH | 1 day prior to treatment start, the superior radiation treatment plan is chosen for treatment delivery
  For each patient, the radiation treatment plan calculated in DIBH and in FB will be compared

SECONDARY OUTCOMES:
Patient compliance defined as 1) patient comfort | Through study completion, an average of 1 month total treatment time
  Patient comfort will be assessed through questionnaires (after first, middle and last treatment fraction) which aim to evaluate the level of information and coaching pre-treatment, the physical treatment environment at the departments, and the health care staff.
Patient compliance defined as 2) breathhold reproducibility | Through study completion, an average of 1 month total treatment time
  Tumor position will be used to evaluate the ability of patients to maintain the breath-hold during the whole course of treatment and to investigate the possibility that patients might get weaker and/or more tired and, thus, unable to perform a stable DIBH as the treatment course progresses. This will be done using the respiratory motion management system.
The accuracy of the treatment delivery | Through study completion, an average of 1 month total treatment time
  Treatment accuracy will evaluated based on daily volumetric imaging, planar kV imaging or surface imaging (e.g. Catalyst, VisionRT). If the tumor is not visible on the planar kV images, the sternum (mediastinal tumors) or the diaphragm (abdominal tumors) will be used as a surrogate structure. If the target position appears reproducible within 5 mm, the patient will be deemed compliant. In addition to the daily online positioning at the treatment machine before each fraction, the reproducibility of the target position will be assessed retrospectively by a medical physicist on a weekly basis.

CONTACTS AND LOCATIONS:
Locations (3):
- Denmark (2):
  - Department of Clinical Oncology, Rigshospitalet, Copenhagen, Danmark
  - Department of Clinical Oncology, Aarhus University Hospital, Aarhus
- Department of Radiation Oncology, Comprehensive Cancer Center, Helsinki University Hospital, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lundgaard AY, Dejanovic D, Berthelsen AK, Andersen FL, Rechner LA, Borgwardt L, Hjalgrim LL, Specht L, Maraldo MV. Baseline FDG PET/CT in free breathing versus deep inspiration breath-hold for pediatric patients with mediastinal lymphoma. Acta Oncol. 2022 Feb;61(2):239-246. doi: 10.1080/0284186X.2021.1974554. Epub 2021 Sep 17. PMID 34533416
- [Derived] Lundgaard AY, Josipovic M, Rechner LA, Bidstrup PE, Hansen R, Damkjaer SS, Joergensen M, Safwat A, Specht L, Hjalgrim LL, Maraldo MV. The Feasibility of Implementing Deep Inspiration Breath-Hold for Pediatric Radiation Therapy. Int J Radiat Oncol Biol Phys. 2020 Apr 1;106(5):977-984. doi: 10.1016/j.ijrobp.2019.12.025. Epub 2020 Jan 28. PMID 32005489
- [Derived] Lundgaard AY, Hjalgrim LL, Rechner LA, Josipovic M, Joergensen M, Aznar MC, Berthelsen AK, Borgwardt L, Johansen C, Loft A, Safwat A, Vaalavirta L, Specht L, Maraldo MV. TEDDI: radiotherapy delivery in deep inspiration for pediatric patients - a NOPHO feasibility study. Radiat Oncol. 2018 Mar 27;13(1):56. doi: 10.1186/s13014-018-1003-4. PMID 29587881